CLINICAL TRIAL: NCT04419922
Title: An Innovative Digital Smoking Cessation Intervention for Low-Income Adults With Substance Use Disorder
Brief Title: A Digital Smoking Cessation Intervention for Adults With Substance Use Disorder
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: BrightView LLC (Industry)
Collaborators: Interact for Health (Unknown); DynamiCare Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 7841-SRezania
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Tobacco Use Disorder; Substance Use Disorders
Keywords: Contingency Management; Smartphone app; Smoking cessation; Tobacco Use Disorder; Tobacco Use Cessation; Nicotine Dependence; Substance Use Disorders
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders; Smoking Cessation; Tobacco Use Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smartphone Contingency Management Arm: 100 participants will be voluntarily recruited at BrightView's Colerain outpatient treatment center to participate in the Smartphone Contingency Management Intervention.
  Interventions: Behavioral: Smartphone Contingency Management Intervention

INTERVENTIONS:
Behavioral: Smartphone Contingency Management Intervention — Participants will provide baseline data on their recent substance use and smoking habits/severity. Participants will 1) download the DynamiCare Rewards app, and 2) receive a Carbon Monoxide breath testing device (iCO™ Smokerlyzer®) and reloadable debit card for receiving financial incentives. Participants will follow instructions on the app to take breath tests and receive incentives if the carbon monoxide breath result is less than 6 ppm (Cessation mode) or lower than 3 of the last 4 tests (Shaping mode). The app will use GPS to track if patients have attended their scheduled BrightView appointments (GPS is not used at any other time) and reward them for all kept appointments. The participant will also be able to view Cognitive Behavioral Therapy (CBT) modules on the app and receive incentives upon completing each module. At all times, the participant retains the right to choose whether to use and when to use the app, device, and funds for a total period of 4 months.
  Other Names: DynamiCare Rewards Intervention; Digital Contingency Management Intervention

SUMMARY:
Adults with substance use disorder (SUD) tend to have started smoking at a younger age and are more likely to be heavy smokers. Due to the many conflicting priorities in this population, smoking cessation is often relegated and ignored by both patients and their healthcare providers. As of 2008, only 2 out of 5 addiction treatment providers in the US offered behavioral treatment for smoking cessation, and less than 1 in 5 offered pharmacotherapy. However, many researchers have found that smoking cessation has positive effects on abstinence from other drugs, as smoking appears to increase craving for and the likelihood of using drugs.

Contingency Management is a highly-effective, evidence based methodology demonstrated to be effective at reducing the use of all types of substances in over 100 randomized controlled trials and 7 meta-analyses. BrightView, an outpatient substance abuse treatment center with several locations across the state of Ohio, has partnered with DynamiCare Health to implement DynamiCare's innovative digital Contingency Management (CM) platform among BrightView's outpatient population of primarily low-income substance use disorder patients with comorbid nicotine dependence/tobacco use disorder.

DynamiCare's platform automates Contingency Management to support smoking cessation interventions via smartphone app. This app rewards participants for negative substance tests and appointment attendance (using GPS tracking) to incentivize abstinence and promote engagement in treatment.

The goal of this study is to reduce tobacco disparities for low-income adult participants using DynamiCare's digital intervention, and to build a rapidly scalable, sustainable process that makes the field of smoking cessation more effective, accountable, and accessible.

DETAILED DESCRIPTION:
In September 2019, the National Institute on Drug Abuse cited research that found smoking rates as high as 85% among patients in treatment for substance use disorder, which is substantially higher than 14% in the general population. Substance use disorder patients tend to start smoking at a younger age and are more likely to be heavy smokers. Due to the many conflicting priorities in this population, smoking cessation is often overlooked and ignored by both patients and their healthcare providers. There are many common misconceptions about comorbid smoking in the substance use disorder population, such as smoking cessation can introduce additional stress that can precipitate relapse. However, this has been proven to be false, as many researchers have found that smoking cessation has positive effects on abstinence from other drugs, as smoking appears to increase craving for and the likelihood of using drugs. In 2018, the National Institute on Drug Abuse cited research that found cigarette smoking increased the likelihood of relapse among people in recovery from substance use disorder. Despite evidence demonstrating the success of concurrent treatment for tobacco and other substances and the positive effects of smoking cessation on substance use outcomes, the substance use disorder population is still systematically undertreated. As of 2008, only 2 out of 5 addiction treatment programs in the US offer behavioral treatment for smoking cessation, and less than 1 in 5 offer pharmacotherapy. Healthcare providers have been urged to do more to help smokers quit. The burden of smoking-related morbidity and mortality in this population is substantial but poorly studied: one study estimated that over half of deaths in patients who recovered from substance use disorder is due to smoking.

While current treatment recommendations include counseling and nicotine replacement therapy, national average annual quit rates remain low at 7%. The quit rate of substance use disorder patients without smoking cessation interventions are as low as 3%, but one meta-analysis found that it increased to 12% with interventions that are incorporated into substance use programs. This demonstrates that strategic investments for this population can induce significant improvements in quit rates. In 2014, the CDC's recommended minimum annual investment for cessation interventions in Ohio was $35.7 million (their ideal investment was $57.7 million)-but the actual expenditures for cessation interventions in Ohio in 2015 were only $7.6 million. Although the expansion of Medicaid under the Affordable Care Act increased coverage for tobacco cessation services nationwide, coverage of tobacco cessation counseling is lagging behind coverage of cessation medications. Barriers to access include copayments and prior authorizations. While the cost-effectiveness of smoking cessation interventions for the substance use disorder population is not well studied, we expect that it is cost-effective because, as mentioned previously, smoking cessation can help improve abstinence, which can further reduce healthcare costs. In addition, concomitant drug use and tobacco use have been found to increase health consequences by 50% compared to drug use and smoking individually.

Current tobacco cessation efforts at BrightView include nicotine replacement therapy and counseling, but quit success rates remain low. Staff are trained to provide patients with the multiple components of medication-assisted treatment (MAT), counseling, and community resources to combat both their addiction(s) and the complex biopsychosocial factors that contribute to them. Despite these resources, tobacco use remains a health problem for the majority patients. Many of them are unemployed and lack reliable transportation, face unstable housing, and have family histories or belong to communities wherein smoking is common and limited cessation services are available.

Contingency Management (CM) is a highly effective, evidence-based methodology. It has been demonstrated to be effective at reducing the use of all types of substances in over 100 randomized controlled trials and 7 meta-analyses. It is often overlooked due to administrative complexities and lack of funding. DynamiCare Health is a multi-service platform, combining software, hardware, and service. It is an innovative technology platform that has automated Contingency Management to support smoking cessation, removing administrative barriers. The DynamiCare app rewards participants for their negative substance and smoking tests to incentivize abstinence and retention in treatment. The app also incentives appointment attendance, using GPS tracking via smartphone. Smoking status is monitored using a pocket-sized carbon monoxide (CO) smokerlyzer.

BrightView and DynamiCare have partnered with Interact for Health to fund and implement a Smartphone Contingency Management Intervention, which seeks to reduce tobacco disparities for low-income adults by providing a successfully tested, evidence-based, innovative digital platform for the treatment of nicotine dependence in participants with substance use disorder. Tobacco abstinence rates will be compared pre- and post- intervention, as well as to the to the national rate quoted in the literature, which is between 7-12%. The goal of the study is to improve abstinence rates to 18%-20%. As a secondary outcome, substance test results will also be evaluated to determine if this smoking cessation intervention had any effect on other substance use behavior.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in a BrightView outpatient substance use disorder program
* Must be active smokers, at least moderate in severity
* Must have substance use disorder as their primary diagnosis
* Must speak and read English adequately to understand smartphone commands and responses
* Must have and use an Android or iOS smartphone with acceptable capability
* Must be willing to participate in breath testing and use of the smartphone

Exclusion Criteria:

* Non-smokers
* Those without a smartphone or access to a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult tobacco smokers with substance use disorder who are currently enrolled in outpatient treatment at BrightView.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence | 4 months
  A comparison of the participant's baseline levels of carbon monoxide to post-intervention levels of carbon monoxide.
Self-Reported Smoker Status | 4 months
  A comparison of the participant's self-reported smoking severity/status pre- and post-intervention.
Attendance Rates | 4 months
  A comparison of the participant's outpatient treatment attendance rates pre- and post-intervention.

SECONDARY OUTCOMES:
Substance Abstinence | 4 months
  A comparison of baseline urine substance test results to post-intervention urine substance test results to measure the impact of smoking cessation on other substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Samin Rezania, PhD, Principal Investigator — Director of Clinical Research
Locations (1):
- BrightView Colerain Addiction Treatment Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Stevens AB, Dorn SB. The State of Tobacco Use Prevention and Cessation in Ohio - Environmental scan and policy implication [Internet]. Ohio: Health Policy Institute of Ohio; 2015 Jun [cited 2019 Oct 19]. (Health Policy Brief). Available from: https://www.philanthropyohio.org/sites/default/files/PolicyBrief_Tobacco.pdf
- [Background] DiGiulio A, Jump Z, Yu A, Babb S, Schecter A, Williams KS, Yembra D, Armour BS. State Medicaid Coverage for Tobacco Cessation Treatments and Barriers to Accessing Treatments - United States, 2015-2017. MMWR Morb Mortal Wkly Rep. 2018 Apr 6;67(13):390-395. doi: 10.15585/mmwr.mm6713a3. PMID 29621205
- [Background] Interact for Health. Tobacco use in Greater Cincinnati. Cincinnati, OH; 2019.
- [Background] Prendergast M, Podus D, Finney J, Greenwell L, Roll J. Contingency management for treatment of substance use disorders: a meta-analysis. Addiction. 2006 Nov;101(11):1546-60. doi: 10.1111/j.1360-0443.2006.01581.x. PMID 17034434
- [Background] Guydish J, Passalacqua E, Tajima B, Chan M, Chun J, Bostrom A. Smoking prevalence in addiction treatment: a review. Nicotine Tob Res. 2011 Jun;13(6):401-11. doi: 10.1093/ntr/ntr048. Epub 2011 Apr 4. PMID 21464202
- [Background] National Institute On Drug Abuse. Tobacco, Nicotine, and E-Cigarettes [Internet]. https://www.drugabuse.gov/publications/research-reports/tobacco-nicotine-e-cigarettes. 2019 [cited 2019 Oct 19]. Available from: https://www.drugabuse.gov/publications/research-reports/tobacco-nicotine-e-cigarettes/introduction
- [Background] CDC. Current Cigarette Smoking Among Adults in the United States [Internet]. Centers for Disease Control and Prevention. 2019 [cited 2019 Oct 19]. Available from: https://www.cdc.gov/tobacco/data_statistics/fact_sheets/adult_data/cig_smoking/index.htm
- [Background] Richter KP, Ahluwalia HK, Mosier MC, Nazir N, Ahluwalia JS. A population-based study of cigarette smoking among illicit drug users in the United States. Addiction. 2002 Jul;97(7):861-9. doi: 10.1046/j.1360-0443.2002.00162.x. PMID 12133125
- [Background] Burling TA, Ramsey TG, Seidner AL, Kondo CS. Issues related to smoking cessation among substance abusers. J Subst Abuse. 1997;9:27-40. doi: 10.1016/s0899-3289(97)90004-3. PMID 9494937
- [Background] Clarke JG, Stein MD, McGarry KA, Gogineni A. Interest in smoking cessation among injection drug users. Am J Addict. 2001 Spring;10(2):159-66. doi: 10.1080/105504901750227804. PMID 11444157
- [Background] de Castro-Neto AG, Rameh-de-Albuquerque RC, de Medeiros PFP, Uchôa R, Santos BS. Neuroscience of Tobacco and Crack Cocaine Use: Metabolism, Effects, and Symptomatology. In: Neuroscience of Nicotine. Elsevier; 2019. p. 403-410.
- [Background] Baca CT, Yahne CE. Smoking cessation during substance abuse treatment: what you need to know. J Subst Abuse Treat. 2009 Mar;36(2):205-19. doi: 10.1016/j.jsat.2008.06.003. Epub 2008 Aug 20. PMID 18715746
- [Background] Epstein DH, Marrone GF, Heishman SJ, Schmittner J, Preston KL. Tobacco, cocaine, and heroin: Craving and use during daily life. Addict Behav. 2010 Apr;35(4):318-24. doi: 10.1016/j.addbeh.2009.11.003. Epub 2009 Nov 12. PMID 19939575
- [Background] Kalman D, Morissette SB, George TP. Co-morbidity of smoking in patients with psychiatric and substance use disorders. Am J Addict. 2005 Mar-Apr;14(2):106-23. doi: 10.1080/10550490590924728. PMID 16019961
- [Background] Mello NK, Mendelson JH, Sellers ML, Kuehnle JC. Effects of heroin self-administration on cigarette smoking. Psychopharmacology (Berl). 1980 Jan;67(1):45-52. doi: 10.1007/BF00427594. PMID 6768078
- [Background] Chait LD, Griffiths RR. Effects of methadone on human cigarette smoking and subjective ratings. J Pharmacol Exp Ther. 1984 Jun;229(3):636-40. PMID 6726650
- [Background] Spiga R, Schmitz J, Day J 2nd. Effects of nicotine on methadone self-administration in humans. Drug Alcohol Depend. 1998 Apr 1;50(2):157-65. doi: 10.1016/s0376-8716(98)00020-9. PMID 9649967
- [Background] Weinberger AH, Platt J, Esan H, Galea S, Erlich D, Goodwin RD. Cigarette Smoking Is Associated With Increased Risk of Substance Use Disorder Relapse: A Nationally Representative, Prospective Longitudinal Investigation. J Clin Psychiatry. 2017 Feb;78(2):e152-e160. doi: 10.4088/JCP.15m10062. PMID 28234432
- [Background] National Institute on Drug Abuse (NIDA). Cigarette Smoking Increases the Likelihood of Drug Use Relapse [Internet]. 2018 [cited 2019 Oct 19]. Available from: https://www.drugabuse.gov/news-events/nida-notes/2018/05/cigarette-smoking-increases-likelihood-drug-use-relapse
- [Background] West R. The clinical significance of "small" effects of smoking cessation treatments. Addiction. 2007 Apr;102(4):506-9. doi: 10.1111/j.1360-0443.2007.01750.x. No abstract available. PMID 17362283
- [Background] Friend KB, Pagano ME. Smoking cessation and alcohol consumption in individuals in treatment for alcohol use disorders. J Addict Dis. 2005;24(2):61-75. doi: 10.1300/J069v24n02_06. PMID 15784524
- [Background] Hughes JR, Kalman D. Do smokers with alcohol problems have more difficulty quitting? Drug Alcohol Depend. 2006 Apr 28;82(2):91-102. doi: 10.1016/j.drugalcdep.2005.08.018. Epub 2005 Sep 26. PMID 16188401
- [Background] Olsen Y, Alford DP, Horton NJ, Saitz R. Addressing smoking cessation in methadone programs. J Addict Dis. 2005;24(2):33-48. doi: 10.1300/J069v24n02_04. PMID 15784522
- [Background] Richter KP, McCool RM, Catley D, Hall M, Ahluwalia JS. Dual pharmacotherapy and motivational interviewing for tobacco dependence among drug treatment patients. J Addict Dis. 2005;24(4):79-90. doi: 10.1300/j069v24n04_06. PMID 16368658
- [Background] Frishman WH. Smoking cessation pharmacotherapy--nicotine and non-nicotine preparations. Prev Cardiol. 2007 Spring;10(2 Suppl 1):10-22. doi: 10.1111/j.1520-037x.2007.05963.x. PMID 17396063
- [Background] Friedmann PD, Jiang L, Richter KP. Cigarette smoking cessation services in outpatient substance abuse treatment programs in the United States. J Subst Abuse Treat. 2008 Mar;34(2):165-72. doi: 10.1016/j.jsat.2007.02.006. Epub 2007 May 23. PMID 17509809
- [Background] Russell MA, Wilson C, Taylor C, Baker CD. Effect of general practitioners' advice against smoking. Br Med J. 1979 Jul 28;2(6184):231-5. doi: 10.1136/bmj.2.6184.231. PMID 476401
- [Background] Gilpin E, Pierce J, Goodman J, Giovino G, Berry C, Burns D. Trends in physicians' giving advice to stop smoking, United States, 1974-87. Tob Control. 1992;1(1):31-36.
- [Background] Schroeder SA. What to do with a patient who smokes. JAMA. 2005 Jul 27;294(4):482-7. doi: 10.1001/jama.294.4.482. PMID 16046655
- [Background] Hurt RD, Offord KP, Croghan IT, Gomez-Dahl L, Kottke TE, Morse RM, Melton LJ 3rd. Mortality following inpatient addictions treatment. Role of tobacco use in a community-based cohort. JAMA. 1996 Apr 10;275(14):1097-103. doi: 10.1001/jama.275.14.1097. PMID 8601929
- [Background] Fiore MC, Smith SS, Jorenby DE, Baker TB. The effectiveness of the nicotine patch for smoking cessation. A meta-analysis. JAMA. 1994 Jun 22-29;271(24):1940-7. PMID 8201739
- [Background] Panel TU and DG. Treating Tobacco Use and Dependence: 2008 Update. US Department of Health and Human Services; 2008.
- [Background] Babb S, Malarcher A, Schauer G, Asman K, Jamal A. Quitting Smoking Among Adults - United States, 2000-2015. MMWR Morb Mortal Wkly Rep. 2017 Jan 6;65(52):1457-1464. doi: 10.15585/mmwr.mm6552a1. PMID 28056007
- [Background] Prochaska JJ, Delucchi K, Hall SM. A meta-analysis of smoking cessation interventions with individuals in substance abuse treatment or recovery. J Consult Clin Psychol. 2004 Dec;72(6):1144-56. doi: 10.1037/0022-006X.72.6.1144. PMID 15612860
- [Background] Bien TH, Burge R. Smoking and drinking: a review of the literature. Int J Addict. 1990 Dec;25(12):1429-54. doi: 10.3109/10826089009056229. PMID 2094682